CLINICAL TRIAL: NCT00520962
Title: New Physiopathogenics Mechanisms Susceptible of Pharmacological Developments (Insulin Resistance and Atherosclerosis)
Brief Title: Screening for Undiagnosed Type 2 Diabetes in New Classes of Subjects at High Risk
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Other Study IDs: 199402-1369/516
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: cardiovascular disease; glucose intolerance; type 2 diabetes; endothelial dysfunction; inflammation; Age> 30 years, male and female; Fasting glucose below 126 mg/dl
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Glucose Intolerance; Inflammation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1,2,3: 1. First degree relatives of patients with type 2 diabetes
  2. Patients with cardiovascular disease and stroke
  3. patients with heart valve disease
- 4: Healthy controls

SUMMARY:
The study aims to evaluate IFG, IGT or unknown type 2 diabetes mellitus in new classes at high risk to develop alterations of glucose metabolism and definition of new pathogenic mechanisms of insulin resistance and atherosclerosis.

The following classes of subjects at high risk will be considered:First degree relatives of patients with type 2 diabetes mellitus, patients with cardiovascular disease and stroke, patients with heart valve disease. age will be > 30 years, both gender.

DETAILED DESCRIPTION:
The primary outcome of the study is evaluation of glucose tolerance, insulin sensitivity and insulin secretion before and 2 hours post-glucose load Secondary outcomes are evaluation of endothelial function, of natriuretic peptides and free fatty acids, and inflammation before and 2 hours post-glucose load. New candidate genes will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Fasting glucose levels <126 mg/dl
* Age >30 years
* Both male and female

Exclusion Criteria:

* Type 1 diabetes
* Known type 2 diabetes mellitus
* Pregnancy
* Impaired kidney and liver function
* Previous history of malignancies

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1997 (Actual)
Dates: Start 1997-06; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PierMarco Piatti, MD, Principal Investigator — IRCSS San Raffaele
Locations (1):
- Medicine Division, Diabetology, Endocrinology and Metabolic Disease Unit, IRCCS San Raffaele, Milan, Italy

REFERENCES:
- [Derived] Monti LD, Lucotti PC, Setola E, Rossodivita A, Pala MG, Galluccio E, LaCanna G, Castiglioni A, Cannoletta M, Meloni C, Zavaroni I, Bosi E, Alfieri O, Piatti PM. Effects of chronic elevation of atrial natriuretic peptide and free fatty acid levels in the induction of type 2 diabetes mellitus and insulin resistance in patients with mitral valve disease. Nutr Metab Cardiovasc Dis. 2012 Jan;22(1):58-65. doi: 10.1016/j.numecd.2010.04.005. Epub 2010 Aug 14. PMID 20709514